CLINICAL TRIAL: NCT02079571
Title: Investigation of Pulse Waves and Channel Entries Produced in Healthy Subjects With Different Constitutions and Their Changes After Treated With Foods of Different Food Attributes
Brief Title: Investigation of Pulse Waves, Channel Entries, and Food Attributes in Healthy Subjects With Different Constitutions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201301076RINB
Record Dates: First submitted 2013-06-13; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Subjects With Different Constitutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- water+ Coconut water (Experimental): forty subjects
  Interventions: Dietary Supplement: Coconut water
- ginger tea +water (Experimental)
  Interventions: Dietary Supplement: ginger tea

INTERVENTIONS:
Dietary Supplement: Coconut water — 250 ml Coconut water for each subject
  Arms: water+ Coconut water
Dietary Supplement: ginger tea — 250 ml for each subject
  Arms: ginger tea +water

SUMMARY:
In traditional Chinese medicine (TCM), hot- and cold-attribute of food ingredients are a major part of dietary therapy. "Eight Principles" including cold/hot, repletion/vacuity, yin/yang and exterior/interior are used for diagnose by Chinese medical doctors. From the perspective of TCM, all constitutions, diseases, herbal medicine and foods can be divided into these two major categories, i.e., cold and hot. Therefore, dietary therapy claims that the attributes of foods should be used to oppose our constitutions in order to harmonize organ functions and maintain human vitality. The true benefit of dietary therapy is considered to be the reestablishment of a harmonious balance between cold and hot, or repletion and vacuity, within the human body.

Previous studies reported that the capillary red blood cell (RBC) velocity in nail fold microcirculation (NFM) of the subjects with hot constitution accelerated significantly after taking the hot attribute aged ginger tea, which might be the result of elevated vagal activity leading to arteriole dilation in these subjects. In contrast, in subjects with cold constitution, capillary RBC velocity decelerated significantly and skin temperature decreased markedly after taking the cold-attribute coconut water, which might have been induced by sympathetic nerve activation causing the arteriole to be constricted. As a result, the use of capillary RBC velocity of NFM measured by laser Doppler anemometer may be a promising way to classify attributes of food ingredients commonly used in Chinese medicine dietary therapy in accordance with different personal constitutions.

Accordingly, it will be a worthwhile task to establish a modern scientific methodology to define the attributes of food ingredients. The aim of this project is to investigate the relationship between food attributes and the physiological signals produced in healthy young subjects with different constitutions. In the first year of this project, investigators are starting to determine the pulse waves produced in healthy subjects with different constitutions by a Smart Pulse Wave Health Evaluation System (S-PULSE). Then, investigators will investigate the relationship between food attributes, channel entries and the physiological signals. Hopefully, the results will have a leverage on the powerful integration capacity within National Taiwan University (NTU) campus to build a hub for global TCM cloud.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult over twenty years old

Exclusion Criteria:

* Severe hypertension
* Cardiovascular diseases

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Determinations of pulse waves and channel entries produced in healthy subjects with different constitutions by a Smart Pulse Wave Health Evaluation System | three hours after each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, MD, Ph D, Study Chair — Chairman and Professor of Primary Care Medicine, College of Medicine, National Taiwan University Hospital
Locations (1):
- Kuan-Hung Lu, Taipei, Taiwan